CLINICAL TRIAL: NCT02831023
Title: Efficacy, Safety, and Pharmacokinetics of Sulphadoxine-pyrimethamine-amodiaquine (SP-AQ), SP-AQ Plus Primaquine, Dihydroartemisinin-piperaquine (DP), DP Plus Methylene Blue for Preventing Transmission of P. Falciparum Gametocytes in Mali
Brief Title: Phase 2 Efficacy Study of Primaquine and Methylene Blue
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Malaria Research and Training Center, Bamako, Mali (Other); Radboud University Medical Center (Other); London School of Hygiene and Tropical Medicine (Other); Heidelberg University (Other); Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UCSF CHR # 15-16839
Record Dates: First submitted 2016-07-06; First posted 2016-07-13 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — fanasil, pyrimethamine drug combination; Primaquine; Methylene Blue; Amodiaquine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- SP-AQ only (Active Comparator): Subjects will receive sulphadoxine-pyrimethamine (SP) as single dose and administered in combination with amodiaquine (AQ), which will be given once daily for 3 days.
  Interventions: Drug: Sulphadoxine-pyrimethamine; Drug: Amodiaquine
- SP-AQ plus PQ (Experimental): Participants in this arm will receive SP-AQ in combination with a single low dose of primaquine at the World Health Organization (WHO) recommended dose of 0.25 mg/kg.
  Interventions: Drug: Sulphadoxine-pyrimethamine; Drug: 0.25 mg/kg primaquine; Drug: Amodiaquine
- DP only (Active Comparator): Participants in this arm will be treated with dihydroartemisinin-piperaquine (DP), which will be administered once a day for three days.
  Interventions: Drug: Dihydroartemisinin-piperaquine
- DP plus MB (Experimental): Study participants in this arm will receive DP as described above combined with once-daily methylene blue (MB) for 3 days, at 15 mg/kg/day (45 mg/kg total over 3 days).
  Interventions: Drug: Methylene blue

INTERVENTIONS:
Drug: Sulphadoxine-pyrimethamine — Each Fansidar tablet is scored containing 500mg sulphadoxine and 25 mg pyrimethamine. Doses will be administered by weight.
  Other Names: Fansidar
  Arms: SP-AQ only; SP-AQ plus PQ
Drug: 0.25 mg/kg primaquine — Primaquine will be administered in an aqueous solution according to weight-based dosing.
  Arms: SP-AQ plus PQ
Drug: Dihydroartemisinin-piperaquine — 160mg/20mg or 320mg/40mg of dihydroartemisinin/piperaquine tablets will be used to administer weight-based doses.
  Other Names: Eurartesim
  Arms: DP only
Drug: Methylene blue — Methylene blue will be given as minitablets in prepackaged sachets according to weight groups.
  Arms: DP plus MB
Drug: Amodiaquine — Amodiaquine will be administered once daily for 3 days, following weight-based dosing of 150 mg tablets.
  Arms: SP-AQ only; SP-AQ plus PQ

SUMMARY:
The purpose of this study is to determine the most efficacious transmission blocking drug regimen for seasonal malaria chemoprophylaxis in Mali. The primary outcome measure will be the proportion of mosquitoes infected pre and post-treatment, assessed through membrane feeding and measured by oocyst prevalence in mosquitoes dissected on day 7 post feed. Primary endpoint will be a within group comparison between the mean of the pretreatment infectivity (Day 0) and infectivity at 7 days post first dose.

DETAILED DESCRIPTION:
Protocol will be shared on request.

ELIGIBILITY:
Inclusion Criteria:

* Glucose-6-phosphate dehydrogenase (G6PD) normal defined by CareStart™ G6PD rapid diagnostic test (RDT) or the OSMMR2000 G6PD semi-qualitative test
* Absence of symptomatic falciparum malaria, defined by fever upon enrollment
* Presence of P. falciparum gametocytes on thick blood film at a density >30 gametocytes/µL (i.e. ≥2 gametocytes recorded in the thick film against 500 white blood cells)
* No allergies to study drugs
* No self-reported use of antimalarial drugs over the past 7 days (as reported by the participant)
* Hemoglobin ≥ 10 g/dL
* Individuals weighing <80 kg
* No evidence of severe or chronic disease
* Written, informed consent

Exclusion Criteria:

* Age < 5 years or > 50 years
* Female gender
* Blood thick film negative for sexual stages of malaria
* Previous reaction to study drugs/known allergy to study drugs
* Signs of severe malaria, including hyperparasitemia, defined as asexual parasitemia > 100,000 parasites / µL)
* Signs of acute or chronic illness, including hepatitis
* Use of other medications (with the exception of paracetamol and/or aspirin)
* Consent not given

Ages: 5 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2016-07; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Mosquito infectivity assessed through membrane feeding assays | 7 day
  Infectivity will be measured by oocyst prevalence in dissected mosquitoes. Primary endpoint will be a comparison between mean of pretreatment infectivity (day 0) and infectivity at days 2 and 7 post first dose.

SECONDARY OUTCOMES:
Gametocyte prevalence, density, and sex ratio measured microscopically and by molecular methods. | 42 days
  Outcome measured at baseline and days 1, 2, 3, 7, 14, 28, and 42 post first dose.
Asexual parasite prevalence and density | 42 days
  Asexual parasitemia will be evaluated by blood smear microscopy and confirmed by more sensitive, molecular methods. Outcome measured at baseline and days 1, 2, 3, 7, 14, 28, and 42 post first dose.
Safety measurements including hemoglobin and signs of hemolysis | 42 days
  The major safety endpoint is hemolysis. For this reason, hemoglobin and methemoglobin values will be measured before treatment, at baseline and on days 1, 2, 3, 7, 14, 28, and 42 post first dose. In addition, clinical review (including additional signs of hemolysis) will be assessed based on active and passive follow-up.
Peak plasma concentration (Cmax) of primaquine | 24 hours
  Outcome measured at hours 1, 2, 4, 6, 8, and 24 post first dose.
Area under the concentration curve (AUC) of primaquine. | 24 hours
  Outcome measured at hours 1, 2, 4, 6, 8, and 24 post first dose.
Elimination half life (t1/2) of primaquine | 24 hours
  Outcome measured at hours 1, 2, 4, 6, 8, and 24 post first dose.
Peak plasma concentration (Cmax) of methylene blue | 24 hours
  Outcome measured at hours 1, 2, 4, 6, 8, and 24 post first dose.
Area under the concentration curve (AUC) of methylene blue | 24 hours
  Outcome measured at hours 1, 2, 4, 6, 8, and 24 post first dose.
Elimination half life (t1/2) of methylene blue | 24 hours
  Outcome measured at hours 1, 2, 4, 6, 8, and 24 post first dose.
Peak plasma concentration (Cmax) of sulphadoxine-pyrimethamine | 24 hours
  Outcome measured at hours 1, 2, 4, 6, 8, and 24 post first dose.
Area under the concentration curve (AUC) of sulphadoxine-pyrimethamine | 24 hours
  Outcome measured at hours 1, 2, 4, 6, 8, and 24 post first dose.
Elimination half-life (t1/2) of sulphadoxine-pyrimethamine | 24 hours
  Outcome measured at hours 1, 2, 4, 6, 8, and 24 post first dose.
Peak plasma concentration (Cmax) of dihydroartemisinin-piperaquine | 24 hours
  Outcome measured at hours 1, 2, 4, 6, 8, and 24 post first dose.
Area under the concentration curve (AUC) of dihydroartemisinin-piperaquine | 24 hours
  Outcome measured at hours 1, 2, 4, 6, 8, and 24 post first dose.
Elimination half-life (t1/2) of dihydroartemisinin-piperaquine | 24 hours
  Outcome measured at hours 1, 2, 4, 6, 8, and 24 post first dose.
Identification of cytochrome P450 (CYP) 2D6 and G6PD polymorphisms | 1 hour
  CYP2D6 and G6PD genotyping will be performed using Thermo Fisher Scientific OpenArray Technology and Copy Number Variation (CNV) assays on the QuantStudio™ 12K Flex Real-Time PCR System.

CONTACTS AND LOCATIONS:
Overall Officials: Roland Gosling, MD, PhD, Principal Investigator — University of California, San Francisco; Alassane Dicko, MD, Principal Investigator — Malaria Research and Training Centre; Teun Bousema, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Malaria Research and Training Centre, Bamako, Mali

IPD SHARING:
Plan to Share IPD: Yes
Data can be shared on request

REFERENCES:
- [Derived] Dicko A, Roh ME, Diawara H, Mahamar A, Soumare HM, Lanke K, Bradley J, Sanogo K, Kone DT, Diarra K, Keita S, Issiaka D, Traore SF, McCulloch C, Stone WJR, Hwang J, Muller O, Brown JM, Srinivasan V, Drakeley C, Gosling R, Chen I, Bousema T. Efficacy and safety of primaquine and methylene blue for prevention of Plasmodium falciparum transmission in Mali: a phase 2, single-blind, randomised controlled trial. Lancet Infect Dis. 2018 Jun;18(6):627-639. doi: 10.1016/S1473-3099(18)30044-6. Epub 2018 Feb 6. PMID 29422384